CLINICAL TRIAL: NCT00958425
Title: Intraoperative Hyaluronic Acid Gel Injection for Improvement of Scar Quality Following Reduction Mammaplasty: a Phase III Double-blinded, Single-centred, Randomized Controlled Study
Brief Title: Intraoperative Hyaluronic Acid Gel Injection for Improvement of Scar Quality Following Reduction Mammaplasty
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Failure of funding
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CDHA-RS/2009-252
Record Dates: First submitted 2009-08-11; First posted 2009-08-13 (Estimated); Last update posted 2024-08-21 (Actual); Status verified 2016-01

CONDITIONS: Cicatrix
MeSH Terms: conditions — Cicatrix

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hyaluronic acid gel (Experimental)
  Interventions: Device: Hyaluronic acid gel
- Saline (Active Comparator)
  Interventions: Device: Saline

INTERVENTIONS:
Device: Hyaluronic acid gel — Hyaluronic acid gel (20 mg/mL), 0.9 mL, intradermal over 2 cm area, once
  Other Names: Prevelle; Restylane; Hyalorunan; Hyaluronate
  Arms: Hyaluronic acid gel
Device: Saline — Normal saline, 0.9 mL, intradermal over 2 cm area, once
  Other Names: Normal saline
  Arms: Saline

SUMMARY:
The purpose of this study is to determine the efficacy of hyaluronic acid gel injections compared to saline injections in improving scar quality in patients undergoing breast reduction surgery. Hyaluronic acid has been implicated in scarless fetal healing, and the investigators therefore hypothesize that injections of hyaluronic acid gel into breast reduction incisions will improve their appearance compared to injections of saline.

ELIGIBILITY:
Inclusion Criteria:

* adequate organ function (BUN < 4.0 mmol/L; serum creatinine < 120 micromol/L; Hgb > 100 g/L; WBC > 4,000/mm3 and < 12,000/mm3; platelets > 100,000/mm3)
* age 18 years or older, with a minimum life expectancy of 2 years
* current non-smoker
* American Society of Anaesthesiology score of 1 or 2
* ability to provide informed consent

Exclusion Criteria:

* previous history of breast surgery; known allergy to polyglactin, poliglecaprone, or injectable hyaluronic acid gel (Restylane or Prevelle)
* history of current or recent (<2 months) immunosuppression
* documented hypersensitivity to streptococcal products
* acute or chronic skin diseases such as folliculitis or psoriasis
* history of bleeding dyscrasia or active anticoagulation (INR>2.0)
* pregnancy or active breast-feeding
* any additional surgical procedures performed in the same surgical session in the same anatomical region
* personal or family history of susceptibility to keloid or hypertrophic scar formation
* Fitzpatrick skin type 5 or 6.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-01-01 (Estimated); Primary Completion 2014-01-01 (Estimated); Study Completion 2014-01-01 (Actual)

PRIMARY OUTCOMES:
Rasch analysis-modified Objective Scar Assessment Score (OSAS) value | 12 months post-operatively

CONTACTS AND LOCATIONS:
Overall Officials: Michael Bezuhly, MD MSc SM FRCSC, Principal Investigator — Capital District Health Authority; Dalhousie University